CLINICAL TRIAL: NCT05697666
Title: The Depth of Neuromuscular Blockade is Not Related to Expiratory Transpulmonary Pressure and Respiratory Mechanics in Moderate to Severe ARDS Patients. A Prospective Cohort Study
Brief Title: Impact of the Depth of Neuromuscular Blockade on Respiratory Mechanics in Moderate to Severe ARDS Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Brieuc (Other)
Responsible Party: Principal Investigator, Nicolas Barbarot, Principal investigator. MD, Intensive Care Unit, Centre Hospitalier de Saint-Brieuc, Centre Hospitalier de Saint-Brieuc
Other Study IDs: 2023-A00165-40
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Distress Syndrome; Ventilator-Induced Lung Injury
Keywords: Oesophageal pressure; Transpulmonary pressure; Train of four; Neuromuscular blockade
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate to severe ARDS adult patients under mechanical ventilation and neuromuscular blockade: no intervention
  Interventions: Other: Modulation of the depth of the neuromuscular blockade

INTERVENTIONS:
Other: Modulation of the depth of the neuromuscular blockade — Analysis of the respiratory mechanics at two times:
  * Facial train of four = 0, indicating a deep neuromuscular blockade
  * Facial train of four > 0, indicating a intermediate to light neuromuscular blockade

SUMMARY:
Neuromuscular blockade (NMB) is proposed in patients with moderate to severe acute respiratory distress syndrome (ARDS). The supposed benefit of these muscle relaxants could be partly linked to their effects on respiratory mechanics by reducing ventilator induced lung injuries (VILI), especially the so called atelectrauma. Although its monitoring is recommended in clinical practice, data about the depth of NMB necessary for an effective relaxation of the thoracic and diaphragmatic muscles and, therefore, the reduction of the chest wall elastance, are scarce. The investigators hypothesised that complete versus partial NMB can modify respiratory mechanics and its partitioning.

DETAILED DESCRIPTION:
The investigators conducted a prospective study to compare the respiratory mechanics of patients with moderate to severe ARDS according to the NMB depth, using an oesophageal pressure catheter (NutriVent®, Sidam) for transpulmonary pressure (PL) assessment, and facial train of four (TOF) for neuromuscular blockade monitoring. The oesophageal balloon was calibrated according to the method recently described to estimate the individual target volume which is assumed to be more adequate. Each patient was analysed at two different times: deep NMB (TOF = 0) and intermediate to light NMB (TOF > 0). The mechanical ventilation parameters were identical for these two measurements. The primary endpoint was the proportion of patients with expiratory transpulmonary pressure (PLexp) greater than or equal to 0 according to the NMB level, in order to assess the risk of region-dependent atelectasis and alveolar opening/closing injury (atelectrauma). Secondary endpoints included: the impact of the depth of NMB on other partition parameters of respiratory mechanics, and the variability of results according to the type of oesophageal balloon calibration.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe ARDS patients with PaO2/FiO2 ratio < 150 mmHg
* Mechanical ventilation, deep sedation and neuromuscular blockade with continuous infusion of cisatracurium for more than 24 hours
* Presence of an oesophageal catheter
* Written informed consent

Exclusion Criteria:

* contraindication of oesophageal catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes mainly pulmonary ARDS with a predominance of SARS-CoV2 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with expiratory transpulmonary pressure greater than or equal to 0 | one day
  Proportion of patients with expiratory transpulmonary pressure greater than or equal to 0 according to the level of neuromuscular blockade (%)

SECONDARY OUTCOMES:
Inspiratory transpulmonary pressure | one day
  Inspiratory transpulmonary pressure according to the level of neuromuscular blockade (cmH20)
Respiratory system compliance | one day
  Respiratory system compliance according to the level of neuromuscular blockade (ml/cmH20)
Chest wall elastance | one day
  Chest wall elastance according to the level of neuromuscular blockade (cmH2O/l)
Pulmonary elastance | one day
  Pulmonary elastance according to the level of neuromuscular blockade (cmH2O/l)
Driving pressure | one day
  Driving pressure according to the level of neuromuscular blockade (cmH20)
Transpulmonary driving pressure | one day
  Transpulmonary driving pressure according to the level of neuromuscular blockade (cmH20)
Plateau pressure | one day
  Plateau pressure according to the level of neuromuscular blockade (cmH20)
Oesophageal balloon calibration | one day
  Proportion of patients with expiratory transpulmonary pressure greater than or equal to 0 according to the oesophageal balloon calibration volume (%)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BARBAROT, MD, Principal Investigator — Centre Hospitalier Saint Brieuc
Locations (1):
- Centre Hospitalier de Saint Brieuc, Saint-Brieuc, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Alhazzani W, Belley-Cote E, Moller MH, Angus DC, Papazian L, Arabi YM, Citerio G, Connolly B, Denehy L, Fox-Robichaud A, Hough CL, Laake JH, Machado FR, Ostermann M, Piraino T, Sharif S, Szczeklik W, Young PJ, Gouskos A, Kiedrowski K, Burns KEA. Neuromuscular blockade in patients with ARDS: a rapid practice guideline. Intensive Care Med. 2020 Nov;46(11):1977-1986. doi: 10.1007/s00134-020-06227-8. Epub 2020 Oct 26. PMID 33104824
- [Background] Guervilly C, Bisbal M, Forel JM, Mechati M, Lehingue S, Bourenne J, Perrin G, Rambaud R, Adda M, Hraiech S, Marchi E, Roch A, Gainnier M, Papazian L. Effects of neuromuscular blockers on transpulmonary pressures in moderate to severe acute respiratory distress syndrome. Intensive Care Med. 2017 Mar;43(3):408-418. doi: 10.1007/s00134-016-4653-4. Epub 2016 Dec 24. PMID 28013329
- [Background] Baedorf Kassis E, Train S, MacNeil B, Loring SH, Talmor D. Monitoring of neuromuscular blockade: a comparison of train-of-four and the Campbell diagram. Intensive Care Med. 2018 Dec;44(12):2305-2306. doi: 10.1007/s00134-018-5420-5. Epub 2018 Oct 22. No abstract available. PMID 30350170